CLINICAL TRIAL: NCT07029737
Title: The SOUND-MCL Study: A Single-arm, Open-label, Multicenter, Phase II Study of Acalabrutinib, in Combination With the R-CHOP Standard of Care, for Previously Untreated Mantle Cell Lymphoma in Spain
Brief Title: A Study to Evaluate Acalabrutinib, in Combination With the R-CHOP Standard of Care, for Previously Untreated Mantle Cell Lymphoma in Spain
Acronym: SOUND-MCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220L00087
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mantle-cell Lymphoma
Keywords: Acalabrutinib; Previously untreated mantle-cell lymphoma; MCL; R-CHOP
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, multicenter, phase II study of acalabrutinib, in combination with the R-CHOP standard of care, for previously untreated mantle cell lymphoma in Spain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Acalabrutinib + R-CHOP standard of care (Induction Phase) plus Acalabrutinib + Rituximab (Maintenance Phase) / Acalabrutinib Monotherapy (Maintenance Phase)
  Interventions: Drug: Acalabrutinib + R-CHOP standard of care; Drug: Acalabrutinib combination with Rituximab; Drug: Acalabrutinib monotherapy

INTERVENTIONS:
Drug: Acalabrutinib + R-CHOP standard of care — Acalabrutinib will be administered 100 mg twice per day (BID) orally (PO) until disease progression if medically appropriate, along with R-CHOP standard of care up to six 21-day cycles of the induction phase.
  Other Names: Induction Phase
Drug: Acalabrutinib combination with Rituximab — If the subject achieves response during the induction phase, acalabrutinib will be administered 100 mg BID PO until disease progression and rituximab 375 mg/m2 on Day 1 of every other 28-day cycle for a maximum of 12 additional doses.
  Other Names: Maintenance Phase
Drug: Acalabrutinib monotherapy — If the subject does not achive response during the induction phase, monotherapy acalabrutinib will be administered 100 mg BID PO until disease progression.
  Other Names: Maintenance Phase

SUMMARY:
This is a single-arm, open-label, multicenter, non-indication seeking phase II trial to describe the efficacy and safety of patients with mantle cell lymphoma (MCL) receiving acalabrutinib in combination with R-CHOP for the front-line treatment of MCL in Spain.

Acalabrutinib will be administered until disease progression if medically appropriate, along with R-CHOP based on institutional standards. After 6 cycles of acalabrutinib in combination with R-CHOP, subjects who tolerate treatment and not progressing, will then receive monotherapy acalabrutinib. In addition, subjects who achieve a response (PR or greater) will receive maintenance rituximab every other 28-day cycle for a maximum of 12 additional doses. Thereafter, subjects receive monotherapy acalabrutinib until disease progression or treatment discontinuation.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, non-indication seeking phase II trial to describe the efficacy and safety of patients with mantle cell lymphoma (MCL) receiving acalabrutinib in combination with the standard of care CIT in Spain, for the front-line treatment of MCL in Spain.

Approximately 55 subjects meeting the eligibility criteria for the study will receive acalabrutinib, in combination with R-CHOP for previously untreated MCL, in approximately 20 Spanish sites.

Acalabrutinib will be administered 100 mg twice per day (BID) orally (PO) until disease progression if medically appropriate, along with R-CHOP based on institutional standards.

A safety run-in will be performed for the first 6 patients older than 75 years included in the study (timeframe: after completing three cycles of the induction phase).

A confirmatory assessment of sufficient efficacy for the acalabrutinib + R-CHOP regimen will be performed for the first 10 patients treated with acalabrutinib + R-CHOP (timeframe: after completing six induction cycles).

After 6 cycles of acalabrutinib in combination with R-CHOP, subjects who tolerate treatment and not progressing, will then receive monotherapy acalabrutinib 100 mg BID. In addition, subjects who achieve a response (PR or greater) will receive maintenance rituximab 375 mg/m2 on Day 1 of every other 28-day cycle for a maximum of 12 additional doses. Thereafter, subjects will receive monotherapy acalabrutinib 100 mg BID (or last tolerated dose) until disease progression or treatment discontinuation for any reason.

The planned duration of recruitment is approximately 12 months. Data will be collected since the inclusion of the first subject, with a maximum prospective follow-up of 30 months since the last subject in. Each subject will be followed up from screening, until the withdrawal from the study, lost to follow-up, death or the end of the study (i.e., 30 months since the last patient in), whichever occurs first.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Adult men or women.
2. Pathologically confirmed MCL, with documentation of chromosome translocation t(11;14)(q13;q32) and/or overexpression of cyclin D1 in association with other relevant markers.
3. MCL requiring treatment and for which no prior systemic anticancer therapies have been received.
4. Unsuitable for autologous stem cell transplantation.
5. Presence of radiologically measurable lymphadenopathy, splenomegaly and/or extranodal lymphoid malignancy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
7. Men who are sexually active and can beget children must agree to use highly effective forms of contraception during the study treatment and for 12 months after the last dose of rituximab or cyclophosphamide, 6 months after the last dose of doxorubicin, 30 days after the last dose of vincristine, and 2 days after the last dose of acalabrutinib, whichever is longest.
8. Men must agree to refrain from sperm donation during the study treatment and for 12 months after the last dose of rituximab or cyclophosphamide, 6 months after the last dose of doxorubicin, 30 days after the last dose of vincristine, and 2 days after the last dose of acalabrutinib, whichever is longest.
9. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing tablets without difficulty.
10. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).
11. WOCBP who are sexually active must use highly effective methods of contraception during the study treatment and for 12 months after the last dose of rituximab or cyclophosphamide, 6 months after the last dose of doxorubicin, 30 days after the last dose of vincristine, and 2 days after the last dose of acalabrutinib, whichever is the longest.
12. Male patients should use barrier contraception from the time of screening until 12 months after the last dose of rituximab or cyclophosphamide, 6 months after the last dose of doxorubicin, 30 days after the last dose of vincristine, and 2 days after the last dose of acalabrutinib, whichever is longest. Male patients wishing to father children in the future should be advised to arrange for the freezing of sperm prior to the start of study treatment.

EXCLUSION CRITERIA:

1. History of prior malignancy except for the following:

   1. Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening and felt to be at low risk for recurrence by treating physician.
   2. Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanomatous skin cancer.
   3. Adequately treated carcinoma in situ without current evidence of disease.
2. Subjects for whom the goal of therapy is tumor debulking before stem cell transplant.
3. Subjects who are deemed by the treating physician to be unfit to tolerate the R-CHOP regimen.
4. Any history of central nervous system (CNS) lymphoma or leptomeningeal disease.
5. Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
6. Major surgical procedure within 28 days before first dose of study drug.
7. Significant cardiovascular disease such as uncontrolled or untreated symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of first dose of study drug, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification at screening. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study.
8. Absolute neutrophil count (ANC) <1.0 x 109/L or platelet count <75 x 109/L; for subjects with disease involvement in the bone marrow, ANC <0.75 x 109/L or platelet count <50 x 109/L. Subjects will only be considered eligible if peripheral blood counts can be maintained independent of growth factors or transfusions during the screening period.
9. Total bilirubin >1.5 x upper limit normal (ULN) unless other reason known; or aspartate aminotransferase (AST) or alanine transaminase (ALT) >2.5 x ULN.
10. Estimated creatinine clearance of <30 mL/min, calculated using the formula of Cockcroft and Gault [(140-age) • mass (kg)/(72 • creatinine mg/dL) • multiply by 0.85 if female].
11. Prothrombin time/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) (in the absence of a lupus anticoagulant) >2.0 x ULN. Exception: Subjects receiving a vitamin K antagonist are excluded; however, those receiving other anticoagulant therapy who have a higher INR/aPTT may be permitted to enroll to this study after discussion with the medical monitor.
12. Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
13. Uncontrolled active systemic fungal, bacterial, viral, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks before first dose of study drug.
14. Known history of infection with human immunodeficiency virus (HIV).
15. Ongoing immunosuppressive therapy, including systemic corticosteroids within 2 weeks before the first dose of study drug.
16. Known history of anaphylaxis or hypersensitivity to any study drug, or any of their components.
17. Serologic status reflecting active hepatitis B or C infection.

    1. Subjects who are anti-HBc positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result before the first dose of study drug. Those who are HbsAg positive or hepatitis B PCR positive will be excluded.
    2. Subjects who are hepatitis C antibody positive will need to have a negative PCR result before the first dose of study drug. Those who are hepatitis C PCR positive will be excluded.
18. Received a live virus vaccination within 28 days of first dose of study drug.
19. History of stroke or intracranial hemorrhage within 6 months of first dose of study drug.
20. History of bleeding diathesis.
21. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before first dose of study drug.
22. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists within 7 days of first dose of study drug.
23. Requires treatment with a strong CYP3A inhibitor/inducer.
24. Concurrent participation in another therapeutic clinical trial.
25. Active cytomegalovirus (CMV) infection (active viremia as evidenced by positive PCR result for CMV DNA).
26. History of confirmed progressive multifocal leukoencephalopathy (PML).
27. Pregnant or breastfeeding women.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (ORR) | From acalabrutinib start to approximately 1 year thereafter
  Investigator-assessed best ORR (CR+PR) as per the Lugano Classification for NHL

SECONDARY OUTCOMES:
Time To Response (TTR) | From acalabrutinib start to the first investigator assessed response; up to 30 months since the last subject in
  TTR, defined as the time from the date of acalabrutinib start to the first investigator-assessed CR or PR per the Lugano Classification for NHL. Measure of interest: median TTR.
Duration of Response (DoR) | From the time of the first documentation of response to disease progression or death; up to 30 months since the last subject in
  DoR, defined as the time from the first documentation of investigator-assessed CR or PR to disease progression per the Lugano Classification for NHL or death from any cause in the absence of disease progression. Measure of interest: 30-month DoR.
Progression-Free Survival (PFS) | From acalabrutinib start to disease progression or death; up to 30 months since the last subject in
  PFS, defined as the time from the date of acalabrutinib start to investigator-assessed disease progression as per the Lugano Classification for NHL or death from any cause, whichever occurs first. Measure of interest: 30-month PFS.
Overall Survival (OS) | From acalabrutinib start to death; up to 30 months since the last subject in
  OS, defined as the time from the date of acalabrutinib start to the date of death from any cause. Measure of interest: 30-month OS.
Safety and tolerability profile | From enrollment to 30 days after the last dose of acalabrutinib or post-acalabrutinib-treatment disease progression; up to 30 months since the last subject in
  Number and percentage of patients with each MedDRA coded and CTCAE graded adverse (AEs) and serious adverse events (SAEs).
  Incidence of AEs of clinical interest for acalabrutinib. Incidence of grade ≥3 AEs. Incidence of AEs leading to acalabrutinib dose modification, temporary interruption or permanent discontinuation.

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Research Site, A Coruña
  - Research Site, Alcorcón
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Donostia / San Sebastian
  - Research Site, Gijón
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Salamanca
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/